CLINICAL TRIAL: NCT05951712
Title: Pre-medication With N-acetylcysteine and Simethicone to Improve Mucosal Visibility During Gastroduodenoscopy: A Double Blind, Randomized Controlled Trial.
Brief Title: Pre-medication With N-acetylcysteine and Simethicone to Improve Mucosal Visibility During Gastroduodenoscopy
Acronym: SIMETHICONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Clinical Professor, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MESE01
Record Dates: First submitted 2023-06-25; First posted 2023-07-19 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Mucosal Erosion
MeSH Terms: interventions — Simethicone; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No Intervention (Placebo Comparator): In this arm, the participants will receive placebo ( 100 ml water) 10-30 minutes before the procedure under the supervision of a trained nurse. All patients will be given standard recommendations before the procedure: at least 8 hours of liquid and solid fasting.
  During endoscopy, mucosal visibility will be evaluated in 6 segments (gastric antrum, lower gastric body, upper gastric body, fundus, first and second part of duodenum), using a scale ranging from 1 to 4 points: (1) no adherent mucus in the gastric mucosa examined; (2) a small amount of mucus in the gastric mucosa examined that does not hinder vision; (3) a large amount of mucus in the gastric mucosa examination, which can be washed thoroughly with <50 mL of water; (4) a large amount of mucus in the gastric mucosa examined which requires ≥50 mL of water for washing.
  Interventions: Other: Placebo
- Simethicone 150 mg (Experimental): In this arm, the participants will receive 150 mg simethicone dissolved in 100 ml water 10-30 minutes before the procedure under the supervision of a trained nurse.All patients will be given standard recommendations before the procedure: at least 8 hours of liquid and solid fasting.
  During endoscopy, mucosal visibility will be evaluated in 6 segments (gastric antrum, lower gastric body, upper gastric body, fundus, first and second part of duodenum), using a scale ranging from 1 to 4 points:(1) no adherent mucus in the gastric mucosa examined; (2) a small amount of mucus in the gastric mucosa examined that does not hinder vision; (3) a large amount of mucus in the gastric mucosa examination, which can be washed thoroughly with <50 mL of water; (4) a large amount of mucus in the gastric mucosa examined which requires ≥50 mL of water for washing.
  Interventions: Drug: Simethicone 150mg
- N Acetyl cysteine 600 mg (Experimental): In this arm the participants will receive 600 mg N-acetyl cysteine dissolved in 100 ml water 10-30 minutes before the procedure under the supervision of a trained nurse.All patients will be given standard recommendations before the procedure: at least 8 hours of liquid and solid fasting.
  During endoscopy, mucosal visibility will be evaluated in 6 segments(gastric antrum, lower gastric body, upper gastric body, fundus, first and second part of duodenum), using a scale ranging from 1 to 4 points:(1) no adherent mucus in the gastric mucosa examined; (2) a small amount of mucus in the gastric mucosa examined that does not hinder vision; (3) a large amount of mucus in the gastric mucosa examination, which can be washed thoroughly with <50 mL of water; (4) a large amount of mucus in the gastric mucosa examined which requires ≥50 mL of water for washing.
  Interventions: Drug: N Acetyl cysteine 600mg
- Simethicone (150 mg) plus N Acetyl cysteine 600 mg combination (Experimental): In this arm, the participants will receive 150 mg simethicone and N-acetyl cysteine dissolved in 100 ml water 10-30 minutes before the procedure under the supervision of a trained nurse.All patients will be given standard recommendations before the procedure: at least 8 hours of liquid and solid fasting.
  During endoscopy, mucosal visibility will be evaluated in 6 segments (gastric antrum, lower gastric body, upper gastric body, fundus, first and second part of duodenum), using a scale ranging from 1 to 4 points:(1) no adherent mucus in the gastric mucosa examined; (2) a small amount of mucus in the gastric mucosa examined that does not hinder vision; (3) a large amount of mucus in the gastric mucosa examination, which can be washed thoroughly with <50 mL of water; (4) a large amount of mucus in the gastric mucosa examined which requires ≥50 mL of water for washing.
  Interventions: Drug: Simethicone 150mg plus N Acetyl cysteine 600 mg

INTERVENTIONS:
Drug: Simethicone 150mg — Impact of simethicone on the mucosal visibility of stomach and duodenum
  Other Names: S
  Arms: Simethicone 150 mg
Drug: N Acetyl cysteine 600mg — Impact of N Acetyl cysteine on the mucosal visibility of stomach and duodenum
  Other Names: NAC
  Arms: N Acetyl cysteine 600 mg
Drug: Simethicone 150mg plus N Acetyl cysteine 600 mg — Impact of simethicone plus N Acetyl cysteine on the mucosal visibility of stomach and duodenum
  Other Names: SPN
  Arms: Simethicone (150 mg) plus N Acetyl cysteine 600 mg combination
Other: Placebo — Impact of water on the mucosal visibility of stomach and duodenum
  Other Names: W
  Arms: No Intervention

SUMMARY:
In this study, we aimed to compare combined premedication with simethicone or N-acetylcysteine (NAC) for mucosal visualisation during esophagogastroduodenoscopy (EGD).

The primary outcome of the study was comparison of total mucosal visibility score (TMVS) between combined pre-medication (Simethicone+ NAC) and individual pre-medication groups (Simethicone and NAC) in patients undergoing EGD. Secondary outcomes included comparison of TMVS between different groups, TMVS in early (10-20 min) versus late (>20-30 min) endoscopy groups, adequate gastric mucosal visibility, detection of lesions and adverse events related to the pre-medications. Adequate and inadequate gastric mucosal visibility was defined as a cumulative score of <7 and ≥7, respectively.

DETAILED DESCRIPTION:
AIM: In this study, we aimed to evaluate the impact of premedication with simethicone or N-acetylcysteine (NAC) for mucosal visualisation during esophagogastroduodenoscopy (EGD).

This is a single-centre, double blinded (patients and endoscopist), randomized trial at a tertiary care academic hospital and approved by institutional review board committee (AIG/IEC-BFI and R 29 /06.2022-04).

The eligibility criteria for enrollment into the study include adult patients (>18 y) undergoing esophagogastroduodenoscopy (EGD). Exclusion criteria for the study are history of upper gastrointestinal surgery, neurological disorder with impaired swallowing, active gastrointestinal bleeding, caustic ingestion, pregnancy, known history of multiple allergies, gastric outlet obstruction, esophageal motility disorders, and contraindication for EGD.

Randomization Patients will be randomly assigned to one of four categories. The randomization algorithm is generated using Random Allocation Software v2.0. Before EGD, a clinical research coordinator will deliver the sealed randomization envelopes to a trained nurse who will administer the solution to the patients after obtaining written informed consent from the study participants. In this trial, both patients and endoscopists will be unaware of the allocation.

Interventions Patients will be randomized to the following 4 groups: group A [100 mL of water (W)]; group B [150 mg simethicone (S)]; group C [600 mg NAC (NAC)]; and group D [150 mg simethicone +600 mg NAC (SPN)]. Patients, nursing staff assisting the procedure, the endoscopist performing the procedure, and the research coordinator collecting the data will be blinded. Identical bottles will be used in all the groups for the purpose of blinding.

A trained nurse not participating in the study will administer the solution 10-30 minutes before EGD. All patients will receive pharyngeal anesthesia with 4 squirts of 10% lidocaine (Xylocaine spray 10%; Neon, Thane, India) before EGD.

After EGD, all patients will be observed for two hours for any immediate adverse events. As feasible, delayed adverse events will be evaluated within 24 hours via telephone inquiry or in-person visits.

Mucosal visibility scoring A pre-defined scoring system will be used for grading mucosal visibility in four regions in stomach (fundus, proximal body, distal body and antrum) and two regions in duodenum [first (D1 and second (D2)]. The mucosal visibility scores range from 1 to 4 (1, no adherent mucus; 2, mild mucus, but not obscuring vision; 3, large amount of mucus obscuring vision, with less than 50 ml water required to clear it; 4, heavy adherent mucus, requiring more than 50 ml water to clear). Total mucosal visibility scores (TMVS) will be estimated by adding individual mucosal visibility scores in six different regions in stomach and duodenum. The TMVS ranges from 6 (best) to 24 (worst) points.

Outcome measures The primary outcome of the study is comparison of TMVS between combined pre-medication (SPN) and individual pre-medication groups (S and NAC) in patients undergoing EGD. Secondary outcomes include comparison of TMVS between different groups (A vs B vs C vs D), TMVS in early (10-20 min) versus late (>20-30 min) endoscopy groups, adequate gastric mucosal visibility, detection of lesions and adverse events related to the pre-medications. Adequate and inadequate gastric mucosal visibility is defined as a cumulative score of <7 and ≥7, respectively.

Sample size calculation In this study we aim to assess the impact of pre-medication on mucosal visibility (MVS) during EGD. We postulated that adequate MV will be at least 15% better in the combined pre-medication (WPSN) arm versus simethicone (WPS) arm.4 The sample size calculated was 346 (173 per group) to demonstrate the superiority of pre-medication with type 1 error as 0.05 and 80% power. Since, the study had four arms the estimated sample size was 692. Considering a 15% drop out rate during the follow-up, the number of cases to be enrolled was calculated to be 796 (199 in each group).

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18-years) capable of giving written, informed consent will be included.
* All eligible subjects undergoing diagnostic endoscopy will be recruited in the study.

Exclusion Criteria:

* History of upperGI tract surgery,
* Gastric cancer
* Need for therapeutic endoscopy and emergency procedures,
* Recent upper GI bleeding
* Caustic ingestion,
* Pregnancy
* Diabetes mellitus
* Asthma
* Allergic reactions to the medications used in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Difference in the proportion of patients with adequate visibility score between the no intervention and the water plus simethicone solution, water plus N Acetyl cysteine solution, water plus simethicone and N Acetyl cysteine solution | 20 minutes
  To achieve adequate mucosal visibility score visibilty score 0 means no mucus in duodenum, stomach

SECONDARY OUTCOMES:
Difference in the proportion of patients with adequate visibility score between the no intervention and the water plus simethicone solution, water plus N Acetyl cysteine solution, water plus simethicone and N Acetyl cysteine solution | 30 minutes
  To achieve adequate mucosal visibility score visibilty score 0 means no mucus in duodenum, stomach

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Dr Nabi, MD, Principal Investigator — ASIAN INSTITUTE OF GASTROENTEROLOGY/AIG HOSPITALS
Locations (1):
- Asian institute of Gastroenterology, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nabi Z, Vamsi M, Goud R, Sayyed M, Basha J, Reddy PM, Reddy R, Reddy P, Manchu C, Darisetty S, Gupta R, Tandan M, Rao GV, Reddy DN. Pre-medication with simethicone and N-acetyl cysteine for improving mucosal visibility during upper gastrointestinal endoscopy: A randomized controlled trial. Indian J Gastroenterol. 2024 Oct;43(5):986-994. doi: 10.1007/s12664-023-01459-0. Epub 2023 Oct 18. PMID 37848768